CLINICAL TRIAL: NCT03505606
Title: Examination of New Visual Acuity and Clinical Crowding Tests for Better Detection of Amblyopia
Brief Title: New Visual Acuity and Crowding Tests for Better Detection of Amblyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FST/FREP/17/739
Record Dates: First submitted 2018-04-04; First posted 2018-04-23 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-08

CONDITIONS: Amblyopia
Keywords: Amblyopia; Visual Acuity; Crowding
MeSH Terms: conditions — Amblyopia; Crowding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Visual acuity tests on control participants
  Interventions: Diagnostic Test: Visual acuity tests
- Strabismic/mixed amblyopes (Experimental): Visual acuity tests on strabismic/mixed amblyopic participants.
  Interventions: Diagnostic Test: Visual acuity tests
- Anisometropic amblyopes (Experimental): Visual acuity tests on anisometropic amblyopic participants.
  Interventions: Diagnostic Test: Visual acuity tests

INTERVENTIONS:
Diagnostic Test: Visual acuity tests — Participants to have visual acuity tested with the three modified vision tests.
  Other Names: Contrast-modulated Cambridge Crowding test; Crowding Distance Test; Enhanced Cambridge Crowding test

SUMMARY:
Amblyopia, or 'lazy eye', is the reduction in vision usually in one eye, due to abnormal visual development without organic cause. It is a preventable and leading cause of monocular vision loss (prevalence of around 3%) and increases lifetime risk of bilateral visual impairment from 10% in the general population, to 18% in amblyopes.

In the UK, vision screening in children aims to detect amblyopia and other undiagnosed visual conditions. Laboratory research suggest that amblyopia could be better detected by modifying standard clinical vision tests to enhance and quantify "crowding". Crowding is the negative effect that surrounding features have on the visibility of a target. Crowding distance and crowding magnitude are considerably greater in amblyopic eyes than in normal healthy eyes. Modifications that should lead to improved amblyopia detection are 1) place letters closer together on a vision chart, 2) define letters by contrast, rather than luminance, and 3) use a new thinner font in the form of numbers, to allow crowding distance in central vision to be measured. In this project, these modifications will be tested in amblyopic children for the first time.

Amblyopic children aged 3 to 11 years (n=32) will be recruited from ACPOS (Addenbrooke's Community Paediatric Ophthalmology Service) at ARU. They will have their vision measured with the three modified tests as well as an uncrowded test. The child will view letters and numbers on a computer screen and respond (verbally or by indicating their choice on a matching card). Testing is fun and game-like with breaks for rewards. Results will be compared to standard vision measurement (SLT: Sonksen LogMAR Test) from the child's ACPOS visit. Amblyopic data will be compared to control data from normal healthy children aged 3 to 11 years (n=200), and age-matched children with normal vision (n=16) from ACPOS (false referrals from school screening).

DETAILED DESCRIPTION:
In the UK, a national vision screening is employed to detect amblyopia and other undiagnosed visual conditions in school-aged children, so that they can be managed effectively. Better detection of amblyopia could be achieved by modifying current visual acuity tests, which measure the spatial resolution limit (or capacity for clarity and sharpness) of vision and by measuring crowding distance; previously unmeasured in a clinical setting. By strengthening crowding magnitude, and better quantifying its spatial distance in paediatric populations, it is hoped that the ability to detect amblyopia, and monitor its improvement with treatment will be significantly enhanced.

Three recent suggestions regarding modifications to current visual acuity tests may lead to improved detection of crowding-sensitive conditions, such as amblyopia. First, closer placement of surrounding letters to the target letter should increase the magnitude of crowding in the amblyopic eye in particular, leading to increased visual acuity differences between eyes. Second, contrast modulated stimuli should enhance crowding in amblyopic eyes. Third, a new thinner font will allow clinical measures of foveal crowding distance. In this project, these three modifications will be tested for the first time in the target clinical population.

Several studies reported that optotypes (letters or symbols) on a vision chart should be placed closer together than they currently are on commercially-available charts, which use 2.5 to 5 stroke-widths separation between target and neighbouring letters. Closer placement disrupts target optotype identification in normal peripheral vision and in central vision of amblyopic eyes due to crowding. In one vision test in the proposed study, a laterally-reversible target letter (e.g., H, O, T or V) will be surrounded by four other letters (U, A, L, C). This arrangement, in which letters were separated by 0.5 optotype widths (or 2.5 stroke widths) was first formally used in the Cambridge Crowding Test. In the proposed experiments, the surrounding letters will be placed 1 stroke-width away from the target letter, the optimal position recommended by recent studies.

Visual acuities for target letters will be measured for both amblyopic and non-amblyopic eyes of child participants, in a clinical environment. These results will be compared with visual acuities acquired during the clinical appointment using the Sonksen logMAR Test (SLT), which is the standard visual acuity test used in Cambridge University Hospital, Addenbrooke's Orthoptic Department

In the Sonksen logMAR Test (SLT), a single line of 4 letters separated from each other by 5 stroke-widths (or 1 optotype width), is contained within a box, separated from the letters also by 5 stroke-widths.

Recognition of target optotypes created by contrast-differences (second-order stimuli) is prone to greater crowding effects than is recognition of optotypes created by luminance-differences (first-order stimuli). This effect is present in normal vision, however even greater visual losses for contrast-defined targets, as well as stronger crowding effects, have been reported in amblyopia. By presenting a contrast-modulated (CM) target letter (H, O, T or V) surrounded by four other letters (U, A, L, C) placed 1 stroke-width away (in the modified Cambridge Crowding Test arrangement), this research aims to examine whether this second-order vision test will exaggerate differences between the eyes of amblyopic children, when compared to those measured in visually 'normal' children. The results will again be compared to those obtained with the Sonksen logMAR test (SLT), a first-order vision test, to compare their sensitivities to amblyopia detection.

Finally, crowding distance, the spatial distance over which crowding occurs, in normal foveal (central) vision is small (2-4 arcmin) and cannot be measured with current standard clinical optotypes due to their large size (5 arcmin for 0.0 logMAR acuity). To get around this difficulty, a new vision test was recently created to quantify the crowding distance or "critical spacing" of crowding . It uses a new "Pelli" font, which is much thinner horizontally than standard clinical fonts, allowing the optotypes to get closer to each other in physical space. This 'Crowding Distance Test' permits quantification of the critical spacing of crowding for the first time in a clinical population. The new "Pelli" font, each optotype appearing like tall skinny numbers, has already been trialled on 'visually normal' school-aged children, but not yet examined on children with greater sensitivity to visual crowding, i.e., amblyopes. The third vision test in the proposed research, will investigate whether or not "crowding distance" measures made in each eye, results in greater inter-ocular differences, leading to better detection of anisometropic and strabismic amblyopia than does the current clinical standard visual acuity test, the Sonksen logMAR test (SLT).

By using closer first-order target optotypes, second-order target optotypes, and quantifying crowding distance in paediatric populations, the ability to detect amblyopia and monitor amblyopia treatment, could be significantly improved for the first time since the 1960s. At that time crowding was first quantified in a clinical population of adult amblyopes and was subsequently incorporated into commercially available tests as best practice.

ELIGIBILITY:
Inclusion Criteria:

* Test participants; Male and female 3 to 11-year-old children diagnosed by ACPOS clinicians as likely having amblyopia (strabismic or anisometropic). They will be tested following 6 weeks (or more) of refractive adaption.
* Control Participants; Male and female 3 to 11-year-old children who have been falsely referred into the Hospital Eye Service (ACPOS) by the visual screening service, but have satisfactory visual functions, as per the national screening guidelines.
* All participants must be able to complete the Sonsken logMAR Test (SLT) either verbally or via use of a matching card.

Exclusion Criteria:

* Uncorrected refractive error.
* The presence of any other vision limiting medical condition, not listed in the inclusion criteria.
* Any prior or existing medical history of epilepsy or seizures.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Waugh, PhD, Study Director — University of Huddersfield
Locations (1):
- Anglia Ruskin University Eye Clinic, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pseudo-anonymised data to be uploaded to ARRO, the university data storage system.

REFERENCES:
- [Background] Chung ST, Li RW, Levi DM. Crowding between first- and second-order letter stimuli in normal foveal and peripheral vision. J Vis. 2007 Mar 9;7(2):10.1-13. doi: 10.1167/7.2.10. PMID 18217825
- [Background] Chung ST, Li RW, Levi DM. Crowding between first- and second-order letters in amblyopia. Vision Res. 2008 Mar;48(6):788-98. doi: 10.1016/j.visres.2007.12.011. Epub 2008 Jan 31. PMID 18241910
- [Background] Danilova MV, Bondarko VM. Foveal contour interactions and crowding effects at the resolution limit of the visual system. J Vis. 2007 Nov 27;7(2):25.1-18. doi: 10.1167/7.2.25. PMID 18217840
- [Background] FLOM MC, WEYMOUTH FW, KAHNEMAN D. VISUAL RESOLUTION AND CONTOUR INTERACTION. J Opt Soc Am. 1963 Sep;53:1026-32. doi: 10.1364/josa.53.001026. No abstract available. PMID 14065335
- [Background] Formankiewicz MA, Waugh SJ. The effects of blur and eccentric viewing on adult acuity for pediatric tests: implications for amblyopia detection. Invest Ophthalmol Vis Sci. 2013 Oct 23;54(10):6934-43. doi: 10.1167/iovs.13-12543. PMID 24071956
- [Background] Hairol MI, Formankiewicz MA, Waugh SJ. Foveal visual acuity is worse and shows stronger contour interaction effects for contrast-modulated than luminance-modulated Cs. Vis Neurosci. 2013 May;30(3):105-20. doi: 10.1017/S0952523813000102. Epub 2013 Apr 25. PMID 23731769
- [Background] Huurneman B, Boonstra FN, Cox RF, Cillessen AH, van Rens G. A systematic review on 'Foveal Crowding' in visually impaired children and perceptual learning as a method to reduce Crowding. BMC Ophthalmol. 2012 Jul 23;12:27. doi: 10.1186/1471-2415-12-27. PMID 22824242
- [Background] Lalor SJH, Formankiewicz MA, Waugh SJ. Crowding and visual acuity measured in adults using paediatric test letters, pictures and symbols. Vision Res. 2016 Apr;121:31-38. doi: 10.1016/j.visres.2016.01.007. Epub 2016 Feb 18. PMID 26878696
- [Background] Siderov J, Waugh SJ, Bedell HE. Foveal contour interaction for low contrast acuity targets. Vision Res. 2013 Jan 25;77:10-3. doi: 10.1016/j.visres.2012.11.008. Epub 2012 Nov 29. PMID 23200866
- [Background] Song S, Levi DM, Pelli DG. A double dissociation of the acuity and crowding limits to letter identification, and the promise of improved visual screening. J Vis. 2014 May 5;14(5):3. doi: 10.1167/14.5.3. PMID 24799622
- [Background] Wong EH, Levi DM, McGraw PV. Is second-order spatial loss in amblyopia explained by the loss of first-order spatial input? Vision Res. 2001 Oct;41(23):2951-60. doi: 10.1016/s0042-6989(01)00189-4. PMID 11704234
- [Background] Wong EH, Levi DM, McGraw PV. Spatial interactions reveal inhibitory cortical networks in human amblyopia. Vision Res. 2005 Oct;45(21):2810-9. doi: 10.1016/j.visres.2005.06.008. PMID 16040080

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Examination of visual acuity using the Sonksen Logmar test (SLT) Examination of Stereoacuity using the Frisby Stereotest and Asteroid Stereotest.
Period: Overall Study
Arm/Group | Control | Strabismic/Mixed Amblyopes | Anisometropic Amblyopes
Started | 25 | 25 | 26
Completed | 24 | 22 | 22
Not Completed | 1 | 3 | 4
Not completed — Unable to complete testing / poor co-operation | 0 | 1 | 0
Not completed — Under observation at Orthoptic clinic for high bilateral hypermetropia | 1 | 0 | 0
Not completed — Stimulus deprivation / previous haemangioma | 0 | 1 | 0
Not completed — Poor compliance with refractive correction | 0 | 0 | 1
Not completed — Insufficient anisometropia | 0 | 0 | 2
Not completed — Ectopia Lentis | 0 | 0 | 1
Not completed — alternation of amblyopic eye | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Strabismic/Mixed Amblyopes | Anisometropic Amblyopes | Total
Number analyzed (Participants) | 24 | 22 | 22 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 22 | 22 | 68
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: Eight participants (1 control and 7 amblyopes) were excluded. The excluded control had high bilateral hypermetropia and had previously been under the observation of an orthoptic department for possible bilateral amblyopia. Seven amblyopes were excluded due to poor compliance with their refractive correction, insufficient anisometropia, Ectopia Lentis, Haemangioma, alternation of amblyopic eye, and non-compliance with testing.
  years | 7.4 [4 to 10] | 7.1 [4 to 10] | 6.2 [3 to 10] | 6.8 [3 to 10]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Eight participants (1 control and 7amblyopes) were excluded. The excluded control had high bilateral hypermetropia and had previously been under the observation of an orthoptic department for possible bilateral amblyopia. Seven amblyopes were excluded due to poor compliance with their refractive correction, insufficient anisometropia, Ectopia Lentis, Haemangioma, alternation of amblyopic eye and non-compliance with testing.
  Participants
    Female | 17 | 9 | 12 | 38
    Male | 7 | 13 | 10 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Eight participants (1 control and 7amblyopes) were excluded. The excluded control had high bilateral hypermetropia and had previously been under the observation of an orthoptic department for possible bilateral amblyopia. Seven amblyopes were excluded due to poor compliance with their refractive correction, insufficient anisometropia, Ectopia Lentis, Haemangioma, alternation of amblyopic eye and non-compliance with testing.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 24 | 22 | 20 | 66
    Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants] — Population: Eight participants (1 control and 7 amblyopes) were excluded. The excluded control had high bilateral hypermetropia and had previously been under the observation of an orthoptic department for possible bilateral amblyopia. Seven amblyopes were excluded due to poor compliance with their refractive correction, insufficient anisometropia, Ectopia Lentis, Haemangioma, alternation of amblyopic eye and non-compliance with testing.
  participants
    United Kingdom | 24 | 22 | 22 | 68
LogMAR visual acuity [Mean (Standard Deviation); unit: logMAR] — Population: Eight participants (1 control and 7 amblyopes) were excluded. The excluded control had high bilateral hypermetropia and had previously been under the observation of an orthoptic department for possible bilateral amblyopia. Seven amblyopes were excluded due to poor compliance with their refractive correction, insufficient anisometropia, Ectopia Lentis, Haemangioma, alternation of amblyopic eye and non-compliance with testing.
  logMAR
    Right eye (controls), amblyopic eye (amblyopes) (SLT) | -0.077 (0.094) | 0.352 (0.231) | 0.195 (0.112) | 0.193 (0.225)
    Left eye (controls), Fellow eye (amblyopes) (SLT) | -0.079 (0.094) | -0.019 (0.083) | -0.032 (0.089) | -0.034 (0.088)

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (LogMAR)
Description: Threshold visual acuity measured in LogMAR
Time Frame: Visual acuities for each participant were measured at a single time point, on a single day; day one of each participants' recruitment.
Population: Eight participants (1 control and 7 amblyopes) were excluded. The excluded control had high bilateral hypermetropia and had previously been under the observation of an orthoptic department for possible bilateral amblyopia. Seven amblyopes were excluded due to poor compliance with their refractive correction, insufficient anisometropia, Ectopia Lentis, Haemangioma, alternation of amblyopic eye and non-compliance with testing.
Measure: Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Control | Strabismic/Mixed Amblyopes | Anisometropic Amblyopes
Number analyzed (Participants) | 24 | 22 | 22
Number analyzed (eyes) | 48 | 44 | 44
logMAR
  Luminance acuity Right eye (control) or Amblyopic eye (amblyopes): number analyzed (eyes) | 24 | 22 | 22
  Luminance acuity Right eye (control) or Amblyopic eye (amblyopes) | 0.004 (0.024) | 0.551 (0.065) | 0.320 (0.025)
  Luminance acuity Left eye (control) or Fellow eye (amblyopes): number analyzed (eyes) | 24 | 22 | 22
  Luminance acuity Left eye (control) or Fellow eye (amblyopes) | 0.005 (0.023) | 0.115 (0.028) | 0.149 (0.022)
  Contrast modulated acuity - Right eye (control) or Amblyopic eye (amblyopes): number analyzed (Participants) | 24 | 21 | 22
  Contrast modulated acuity - Right eye (control) or Amblyopic eye (amblyopes): number analyzed (eyes) | 24 | 21 | 22
  Contrast modulated acuity - Right eye (control) or Amblyopic eye (amblyopes) | 0.361 (0.023) | 0.836 (0.050) | 0.676 (0.028)
  Contrast modulated acuity - Left eye (controls) or Fellow eye (amblyopes): number analyzed (Participants) | 24 | 21 | 22
  Contrast modulated acuity - Left eye (controls) or Fellow eye (amblyopes): number analyzed (eyes) | 24 | 21 | 22
  Contrast modulated acuity - Left eye (controls) or Fellow eye (amblyopes) | 0.358 (0.021) | 0.470 (0.026) | 0.479 (0.023)

2. Primary Outcome: Foveal Crowding Distance (Degrees)
Description: Foveal critical crowding distance measured in degrees
Time Frame: Crowding distances for each participant were measured at a single time point, on a single day; day one of each participants' recruitment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Degrees
Units Other Than Participants: eyes
Arm/Group | Control | Strabismic/Mixed Amblyopes | Anisometropic Amblyopes
Number analyzed (Participants) | 24 | 22 | 22
Number analyzed (eyes) | 48 | 44 | 44
Degrees
  Foveal crowding distance Trigram format- Right eye (controls) and Amblyopic eye (amblyopes): number analyzed (Participants) | 24 | 21 | 22
  Foveal crowding distance Trigram format- Right eye (controls) and Amblyopic eye (amblyopes): number analyzed (eyes) | 24 | 21 | 22
  Foveal crowding distance Trigram format- Right eye (controls) and Amblyopic eye (amblyopes) | 0.088 (0.008) | 0.501 (0.144) | 0.197 (0.014)
  Foveal crowding distance repeated format - Right eye (controls) and Amblyopic eye (amblyopes): number analyzed (Participants) | 24 | 21 | 22
  Foveal crowding distance repeated format - Right eye (controls) and Amblyopic eye (amblyopes): number analyzed (eyes) | 24 | 21 | 22
  Foveal crowding distance repeated format - Right eye (controls) and Amblyopic eye (amblyopes) | 0.096 (0.011) | 0.561 (0.122) | 0.225 (0.025)
  Foveal crowding distance trigram format - Left eye (controls) and Fellow eye (amblyopes): number analyzed (Participants) | 24 | 21 | 22
  Foveal crowding distance trigram format - Left eye (controls) and Fellow eye (amblyopes): number analyzed (eyes) | 24 | 21 | 22
  Foveal crowding distance trigram format - Left eye (controls) and Fellow eye (amblyopes) | 0.088 (0.008) | 0.106 (0.008) | 0.110 (0.009)
  Foveal crowding distance repeated format - Left eye (controls) and Fellow eye (amblyopes): number analyzed (Participants) | 24 | 21 | 22
  Foveal crowding distance repeated format - Left eye (controls) and Fellow eye (amblyopes): number analyzed (eyes) | 24 | 21 | 22
  Foveal crowding distance repeated format - Left eye (controls) and Fellow eye (amblyopes) | 0.103 (0.004) | 0.113 (0.007) | 0.120 (0.009)

ADVERSE EVENTS:
Time Frame: Each participant was assessed on a single day, so 1 day.
Arm/Group | Control | Strabismic/Mixed Amblyopes | Anisometropic Amblyopes
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/26

LIMITATIONS AND CAVEATS:
Delays with recruitment and testing due to COVID-19 lockdowns

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT03505606/Prot_SAP_ICF_000.pdf